CLINICAL TRIAL: NCT06262737
Title: Single-center Study Measuring OSDI Dry Eye Score in Patients Undergoing an Anti-VEGF Induction Protocol
Acronym: PISO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RBHP 2023 CHIAMBARETTA; 2023-A01121-44 (Registry Identifier: ANSM)
Record Dates: First submitted 2023-10-17; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-10

CONDITIONS: Macular Degeneration; Diabetic Macular Edema; Retinal Vein Occlusion
MeSH Terms: conditions — Macular Degeneration; Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess the sensation of ocular dry eye symptom after an intravitreal injection of anti-VEGF.

DETAILED DESCRIPTION:
The recrutement of the patient is done during the inclusion of the patient by the nurses of the ophtalmological service of clermont-ferrand and confirm by an ophtalmologist of the service.

A mesure of the OSDI is done before the injection, then at 1 day, on week by a phone call. Each of this mesures are done for the 2 other injections.

Before each of this injection, a clinical mesure is done by a lacrydiag: the atrophy of the meibomian glands, the non-invasive break-up time, interferometry, the heigh of the tear meniscum.

ELIGIBILITY:
Inclusion Criteria:

* Patient with exsudative age-related macular degeneration, diabetic macular edema or retinal vein occlusion
* Patient with 3 ocular intravitreal injections of anti-VEGF in one eye

Exclusion Criteria:

* pregnant or breastfeeding woman
* intravitreal injection before the study
* intravitreal injection in both eyes
* allergy of betadine
* guardianship patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with retinal injury who will have 3 injections as the induction protocol (1 injection per month) for one eye and that didn't had any injection before.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
OSDI | before the injection and at 1 day
  Ocular Surface Disease Index: 12 questions treating of either the sensation, the visual impact and the environemental impact of the dry eye disease

SECONDARY OUTCOMES:
OSDI | before the injection and at 1 week
  Ocular Surface Disease Index: 12 questions treating of either the sensation, the visual impact and the environemental impact of the dry eye disease
HM | before each injection
  MH: hauteur méniscal : high of meniscal tear film
AM | before each injection
  Atrophie meibomienne: meibomian atrophy
NIBUT 1 | before each injection
  First Non Invasive Break-Up Time: time when the tear film lose is regularity regardless of is location
NIBUT 2 | before each injection
  Average Non Invasive Break-Up Time : average time when the tear film lose is regularity for each location
Interferometry | before each injection
  Interferometry: High of the lipid film of the tear

CONTACTS AND LOCATIONS:
Overall Officials: Frederic CHIAMBARETTA, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France